CLINICAL TRIAL: NCT04582123
Title: The Comparison of Cross Pin Configurations in the Treatment of Gartland Type III Supracondylar Humerus Fractures: 2 Pins Versus 3 Pins
Brief Title: Comparison of Cross Pin Configurations in Supracondylar Humerus Fracture Treatment: 2 Pins Versus 3 Pins
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2014/250
Record Dates: First submitted 2020-10-05; First posted 2020-10-09 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Supracondylar Humerus Fracture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- comparison of two cross pin fixation methods (Other): Fixation of supracondylar humerus fractures with 2 crossed pins and 3 crossed pins are compared in terms of Flynn's criteria
  Interventions: Procedure: crossed pin configuration

INTERVENTIONS:
Procedure: crossed pin configuration — comparison of two crossed pin fixation methods

SUMMARY:
The objective of this prospective randomized controlled trial is to evaluate and compare the outcome of the 2wire vs 3 wire crossed pin configurations in the management of supracondylar humeral fractures in children.

DETAILED DESCRIPTION:
Fortyfive children with supracondylar humeral fractures were randomly divided into two groups. One group was treated with 2 crossed pins and the other group with 3 crossed pins. The mean age was 6.04±2.49 (1-12).. The follow-up period was 5 years, with no patients lost to follow up.

Intervention: Twentytwo patients were managed by 2 crossed and 23 by 3 crossed pin method. All surgeries were performed by the same surgeon.

Main Outcome Measurements: Postoperative stability, ulnar nerve injury, range of motions, and pin tract infections were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria was children with closed extension Type III of supracondylar fracture of humerus.

Exclusion Criteria:

* Patients with Type I and Type II injuries, flexion type injuries, open fractures and patients above the age of 12 years were excluded from the study.

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2015-01-15 (Actual); Primary Completion 2020-01-24 (Actual); Study Completion 2020-01-24 (Actual)

PRIMARY OUTCOMES:
functional outcome of two fixation techniques | 5 years
  comparison of Flynn's criteria